CLINICAL TRIAL: NCT00563641
Title: Very Early Surfactant Without Mandatory Ventilation In Premature Infants Treated With Early Continuous Positive Airway Pressure-A Randomized Controlled Trial
Brief Title: Very Early Surfactant and NCPAP for Premature Infants With RDS
Acronym: CNRNCPAP
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Colombian Neonatal Research Network (Other)
Collaborators: Pontificia Universidad Javeriana (Other); Vanderbilt University School of Medicine (Other); Abbott (Industry); Fisher and Paykel Healthcare (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ColombianCNRNCPAP trial; Abbott Laboratories Grant
Record Dates: First submitted 2007-11-23; First posted 2007-11-26 (Estimated); Last update posted 2007-11-26 (Estimated); Status verified 2007-11

CONDITIONS: Respiratory Distress Syndrome; Pneumothorax/Pulmonary Intersticial Emphysema; Chronic Lung Disease
Keywords: NCPAP; Very early surfactant
MeSH Terms: conditions — Respiratory Distress Syndrome; Pneumothorax

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): Early NCPAP plus very early surfactant
  Interventions: Other: Very early surfactant and bubble NCPAP
- 2 (Active Comparator): NCPAP alone
  Interventions: Other: bubble NCPAP

INTERVENTIONS:
Other: Very early surfactant and bubble NCPAP — For patients randomized to early NCPAP plus surfactant, 4ml/kg of surfactant were administered through an endotracheal tube in two aliquots, 2 minutes apart followed by positive pressure ventilation administered for one minute with a Neopuff Infant Resuscitator pre-set to give a peak pressure of 20 cm H2O and 5 cm H2O of positive end expiratory pressure. Infant was then extubated and placed on NCPAP of 6 cmH2O
  Arms: 1
Other: bubble NCPAP — Premature infants randomized to bubble NCPAP alone will continue on NCPAP until they reach "yes or no" treatment failure criteria.
  Arms: 2

SUMMARY:
The present study will test the use of very early nasal continuous airway pressure(NCPAP)with and without surfactant in premature infants with clinical evidence or respiratory distress syndrome. We hypothesize that premature infants exposed to very early NCPAP and surfactant will require less mechanical ventilation compared to those premature infants exposed to NCPAP alone.

DETAILED DESCRIPTION:
Premature infants who are not intubated during the first 15 minutes of life and who develop clinical evidence of respiratory distress or need for oxygen requirement between 15 and 60 minutes of life, will be placed on bubble NCPAP of 6 cm H2O. Randomization envelops will them be opened and patients will be assigned to continuation on NCPAP alone (Control Group) or to NCPAP plus very early surfactant therapy (Treatment Group). Patients assigned to the treatment group will be transiently intubated for surfactant administration, extubated, and placed back on NCPAP of 6 cm H2O. Both groups will then be followed over time to determine which infants meet treatment failure criteria defined as: Treatment failure was defined a priori by either failure of adequate oxygenation or ventilation as follows: "1" FiO2 greater than 0.75 for more than 30 minutes to maintain SpO2 within the pre-established target ranges, "2" persistent or recurrent desaturation below 80% that did not respond to suctioning of the airways and PPV, "3" PCO2>65 mmHg and pH<7.22 on an arterial or capillary blood gas analysis, in association with increased work of breathing. Infants in the Treatment Group who cannot be extubated after their initial dose of surfactant because of clinical instability will be analyzed as treatment failures. Premature infants that meet treatment failure criteria on either arm will be intubated and placed on mechanical ventilation and given surfactant rescue doses according to the criteria of the participating institutions. Premature infants with respiratory distress syndrome who do not meet treatment failure criteria in both groups will remain on NCPAP until their respiratory failure improves.

ELIGIBILITY:
Inclusion Criteria:

* Gestational age of 27 to 31 6/7 weeks,
* Postnatal age between 15 and 60 minutes,
* Supplemental oxygen requirement or evidence of increased work of breathing (tachypnea, intercostal retractions, nasal flaring, or grunting), and
* Prenatal consent.

Exclusion Criteria:

* Apgar score less than 2 at 5 minutes,
* Intubation prior to randomization,
* Prenatal diagnosis of major congenital anomalies,
* Prolonged rupture of membranes of greater than 3 weeks duration, and
* Infants who were likely to be transferred to another center soon after birth were not enrolled in the study.

Ages: 27 Weeks to 31 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 278 (Actual)
Dates: Start 2004-01; Study Completion 2006-12 (Actual)

PRIMARY OUTCOMES:
Need for mechanical ventilation | Death or discharge from the NICU

SECONDARY OUTCOMES:
Neonatal mortality | During hospitalization in the NICU
Air leak syndrome | death or discharge from the NICU
Oxygen dependency at 36 weeks post menstrual age | Death or discharge from the NICU

CONTACTS AND LOCATIONS:
Overall Officials: Mario A Rojas, MD, MPH, Principal Investigator — Vanderbilt University
Locations (1):
- Department of Epidemiology and Biostatistics Pontificia Universidad Javeriana, Bogota, Cundinamarca, Colombia

REFERENCES:
- [Background] Rojas MA, Lozano JM, Rojas MX; Colombian Neonatal Research Network. International collaborative research: a Colombian model that promotes infant health and research capacity. J Perinatol. 2007 Dec;27(12):738-43. doi: 10.1038/sj.jp.7211827. Epub 2007 Sep 20. PMID 17882265
- [Derived] Rojas MA, Lozano JM, Rojas MX, Laughon M, Bose CL, Rondon MA, Charry L, Bastidas JA, Perez LA, Rojas C, Ovalle O, Celis LA, Garcia-Harker J, Jaramillo ML; Colombian Neonatal Research Network. Very early surfactant without mandatory ventilation in premature infants treated with early continuous positive airway pressure: a randomized, controlled trial. Pediatrics. 2009 Jan;123(1):137-42. doi: 10.1542/peds.2007-3501. PMID 19117872